CLINICAL TRIAL: NCT07177417
Title: EVax-3: Human Upper and Lower Airway Mucosal Immune Response to FluMist Vaccination
Brief Title: Characterizing the Human Airway Immune Response to FluMist Vaccination
Acronym: EVax-3
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Philip Mudd, Assistant Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202505085
Record Dates: First submitted 2025-09-09; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Healthy Young Adults; Influenza Vaccines; Influenza Vaccine Response
Keywords: FluMist; bronchoscopy; bronchoalveolar lavage; endobronchial biopsy; nasopharyngeal swab; inactivated influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — FluMist; fluarix; Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- FluMist bronchoscopy group (Experimental): Individuals who undergo all bronchoscopy procedures randomized to receive FluMist vaccine
  Interventions: Biological: FluMist; Procedure: bronchoscopy
- FluMist no bronchoscopy group (Experimental): Individuals who do not complete day 14 or day 90 bronchoscopy procedures randomized to receive FluMist vaccine
  Interventions: Biological: FluMist
- inactivated influenza vaccine bronchoscopy group (Active Comparator): Individuals who undergo all bronchoscopy procedures randomized to receive inactivated influenza vaccine
  Interventions: Biological: inactivated influenza vaccine; Procedure: bronchoscopy
- inactivated influenza vaccine no bronchoscopy group (Active Comparator): Individuals who do not complete day 14 or day 90 bronchoscopy procedures randomized to receive inactivated influenza vaccine
  Interventions: Biological: inactivated influenza vaccine

INTERVENTIONS:
Biological: FluMist — intranasal administered live attenuated influenza vaccine
  Arms: FluMist bronchoscopy group; FluMist no bronchoscopy group
Biological: inactivated influenza vaccine — intramuscular administered inactivated influenza vaccine
  Other Names: FLUARIX
  Arms: inactivated influenza vaccine bronchoscopy group; inactivated influenza vaccine no bronchoscopy group
Procedure: bronchoscopy — bronchoscopy with bronchoalveolar lavage and endobronchial biopsy sampling
  Arms: FluMist bronchoscopy group; inactivated influenza vaccine bronchoscopy group

SUMMARY:
The goal of this clinical trial is to measure the immune response in the blood, nose, and lungs after participants receive either the FDA-approved inactivated influenza vaccine or the FDA-approved intranasal FluMist vaccine. The study will evaluate immune responses in groups of healthy, non-pregnant, volunteers between the ages of 18 and 40. The main purpose of the study is to measure the change in influenza vaccine-specific antibodies in the lower lungs and nose between vaccination and 14 days after participants receive the vaccine. All participants will be randomized to receive one of the two seasonal flu vaccines and will have blood and back of the nose swabs collected throughout the study. Some study participants will choose to undergo optional bronchoscopy procedures and will be included in the part of the study looking at lower lung immune responses.

DETAILED DESCRIPTION:
Study Design/Methodology: Prospective randomized controlled trial; Study Duration: 2 years; Number of Subjects: 30; Subject Participation Duration: 4 months; Description of Interventions: Eligible healthy participants who have not received a seasonal influenza vaccine within the past 9 months will complete written informed consent. Enrolled participants will be randomized to receive either an FDA-approved intramuscular seasonal egg-based inactivated influenza vaccine (IIV) (N=15) or the FDA-approved seasonal FluMist intranasal live attenuated influenza vaccine (N=15) on study day 0. Blood samples and nasopharyngeal swabs will be collected at the time of study enrollment (up to 45 days prior to vaccination) and on days 3±1, 7±2, 14±3, 28±5, and 90±14 post-vaccination. Sixteen participants (N=8 in each vaccine group) will be enrolled for optional research bronchoscopy procedures. Research bronchoscopies will include bronchoalveolar lavage (BAL) and endobronchial biopsy (EBBx) sample collection. Research bronchoscopies will be performed prior to vaccination and on study days 14±3 and 90±14. Screening safety laboratory studies and screening chest x-ray imaging will be performed on subjects undergoing research bronchoscopies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-40 years
* Able to understand and give written informed consent
* In stable health, as determined by medical history and targeted physical exam related to the history

Exclusion Criteria:

* Prisoners
* Anyone unable to provide full written informed consent
* Pregnant women and nursing mothers or women who are planning to become pregnant during the study interval
* Female subjects who are sexually active with male partners who are not actively on hormonal contraception or who do not have an IUD in place
* Vaccination with a seasonal influenza vaccine or documented infection with seasonal influenza in the past 9 months
* Receipt of any vaccine in the 28 days prior to the pre-vaccination study visit or planned receipt of any non-study vaccine before completion of study day 28 visit
* Current smokers
* BMI > 40
* Individuals with an immunocompromising medical condition or who have received systemic immunosuppressants or immune-modifying drugs for > 14 days in total within 6 months prior to screening (for corticosteroids ≥ 10 mg/day of prednisone equivalent for > 14 days total) or is anticipating the need for immunosuppressive treatment at any time during participation in the study
* Individuals who currently have symptomatic acute or unstable chronic disease requiring medical or surgical care, to include significant change in therapy or hospitalization, at the discretion of the investigator
* History of excessive alcohol consumption, drug abuse, psychiatric conditions, social conditions or occupational conditions that in the opinion of the investigator would preclude compliance with the study
* Have donated blood, blood products, or bone marrow within 30 days before study entry, plan to donate blood at any time during the duration of study participation, or plan to donate blood within 30 days after the last blood draw.
* Current ongoing participation in a clinical trial evaluating an investigational agent unless the trial is in follow up only and the last dose of the investigational agent was taken >30 days or >5 half-lives prior to enrollment, whichever is greater.
* Any condition in the opinion of the investigator that would interfere with the proper conduct of the trial.

For participants willing to undergo bronchoscopy:

* Any known chronic pulmonary, cardiovascular, neurologic or hematologic disorder that could, in the opinion of the physician bronchoscopist or the principal investigator, put the subject at unnecessary risk from the sedation and bronchoscopy procedures. These conditions may include, but are not limited to, the following: asthma, COPD, obstructive sleep apnea, pulmonary fibrosis, cystic fibrosis, pulmonary hypertension, heart failure, previous myocardial infarction, hypertrophic cardiomyopathy, supraventricular tachycardia, paraplegia, quadriplegia, epilepsy, sickle cell disease, hemophilia, chronic anemia or active cancer.
* Coagulopathy (primary or iatrogenic) which would contraindicate bronchoscopy for participants willing to have those procedures done. Any participant with an INR>1.4, PTT>40 or platelet count <100,000 at study screening will not be eligible for bronchoscopy.
* Evidence of significant pulmonary disease on the day of bronchoscopy, including pulse oximetry with oxygen saturation of 92% or less on room air, or infiltrate or pleural effusion on an upright PA and lateral chest x-ray performed on the day of bronchoscopy.
* Allergy or contraindication to anesthesia for participants willing to have bronchoscopy done.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Change in vaccine-specific mucosal antibody response following vaccination | From samples before vaccination and day 14 after vaccination.
  Measure the change in influenza vaccine strain-specific hemagglutinin and neuraminidase antibody titers found at the upper and lower airway mucosal surface between day 0 and day 14 after administration of FluMist intranasal influenza vaccination versus standard dose trivalent IIV using ELISA.

SECONDARY OUTCOMES:
Change in vaccine-specific circulating antibody following vaccination. | From samples before vaccination and day 14 after vaccination.
  Measure the change in influenza vaccine strain-specific antibody titers found in blood between day 0 and day 14 after administration of FluMist intranasal influenza vaccination versus standard dose IIV using ELISA.
Change in influenza-specific mucosal and circulating CD8+ T cells following vaccination. | From samples before vaccination and day 14 after vaccination.
  Measure the change in the magnitude of influenza-specific CD8+ T cells found in the blood, the nasopharynx, the lower airways and the lung tissue between day 0 and day 14 using flow cytometry with influenza-specific HLA class I tetramer reagents.
Change in influenza-specific mucosal and circulating B cells following vaccination. | From samples before vaccination and day 14 after vaccination.
  Measure the change in the magnitude of influenza-specific B cells found in the blood and the lung tissue between day 0 and day 14 using flow cytometry with influenza strain-specific fluorescently-labeled HA probes.
Change in vaccine-specific mucosal antibody response 3 months after vaccination | From samples taken on day 14 after vaccination and day 90 after vaccination.
  Measure the change in influenza vaccine strain-specific antibody titers found at the lower airway mucosal surface and at the nasopharyngeal mucosal surface between day 14 and day 90 using ELISA.
Change in influenza-specific mucosal and circulating CD8+ T cells and B cells 3 months after vaccination. | From samples taken on day 14 after vaccination and day 90 after vaccination.
  Measure the change in the magnitude of influenza-specific CD8+ T cells and B cells found in the blood, the nasopharynx, the lower airways and the lung tissue between day 14 and day 90 using flow cytometry with influenza-specific HLA class I tetramer reagents and strain-specific fluorescently-labeled HA probes.

CONTACTS AND LOCATIONS:
Overall Officials: Philip A. Mudd, M.D., Ph.D., Principal Investigator — Washington University in Saint Louis School of Medicine
Locations (1):
- Washington University in Saint Louis School of Medicine Emergency Care and Research Core, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No